CLINICAL TRIAL: NCT06366243
Title: A Phase 1, Open-Label, Fixed-Sequence Trial to Evaluate the Effect of Esomeprazole and Gastric pH-Altering on the Pharmacokinetics of Emraclidine in Healthy Adult Participants
Brief Title: A Trial to Evaluate the Effect of Esomeprazole on the Pharmacokinetics of Emraclidine in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-HV-1012
Record Dates: First submitted 2024-04-11; First posted 2024-04-15 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emraclidine 30 mg + Esomeprazole 40 mg (Experimental): Participants will receive a single oral dose of 30 milligrams (mg) emraclidine on Day 1 of Treatment Period 1. After 6 days following the single dose of emraclidine in Treatment Period 1, participants will receive 40 mg esomeprazole, orally, once daily (QD) on Days 1 to 5 of Treatment Period 2. On Day 6 of Period 2, participants will receive 40 mg esomeprazole followed by a single oral dose of 30 mg emraclidine.
  Interventions: Drug: Emraclidine; Drug: Esomeprazole

INTERVENTIONS:
Drug: Emraclidine — Oral tablet
  Other Names: CVL-231
Drug: Esomeprazole — Oral delayed-release capsule
  Other Names: Nexium

SUMMARY:
The primary purpose of this study is to evaluate the potential of gastric pH-dependent drug-drug interaction effect of esomeprazole, a proton pump inhibitor (PPI), on the pharmacokinetics (PK) of emraclidine in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women of childbearing potential must agree to use at least a highly effective birth control method, during the trial and for 7 days after the last dose of investigational medicinal product (IMP).
* Body mass index of 18.5 to 35.0 kilogram per meter square (kg/m2), inclusive, and a total body weight ≥50 kg (110 [pounds] lbs).
* Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECGs, vital sign measurements, and laboratory test results, as evaluated by the investigator.

Exclusion Criteria:

* Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
* "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

  * Suicidal Ideation Item 3 (Active Suicidal Ideation with Any Methods [Not Plan] without Intent to Act)
  * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
  * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent)
  * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior)
* "Yes" responses for any of the following items on the C-SSRS (within past 12 months):

  * Suicidal Ideation Item 1 (Wish to be Dead)
  * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts)
* Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
* Use of any prescription and over-the-counter medications from 28 days prior to first dose of IMP or likely to require concomitant therapy. Vaccinations or boosters within 28 days of planned dosing or while on trial are prohibited.
* Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B total core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
* Positive drug screen (including cotinine and tetrahydrocannabinol [THC]) or a positive test for alcohol.
* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement, if deemed necessary:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2× upper limit of normal (ULN).
  * Total bilirubin >1.5×ULN. If Gilbert's syndrome is suspected, total bilirubin >1.5×ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.
* Known allergy or hypersensitivity to the IMP, closely related compounds, or any of their specified ingredients.
* Female participants who are pregnant, breastfeeding, or planning to become pregnant during IMP treatment or within 7 days after the last dose of IMP. Women of childbearing potential must have a negative serum pregnancy test result at the Screening Visit and a negative urine pregnancy test result at Check-in.
* Received IMP in a clinical trial of emraclidine.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Emraclidine | Pre-dose and at multiple time points post-dose on Days 1 to 6 in Period 1 and Days 6 to 11 in Period 2
Time to Maximum (Peak) Plasma Concentration (Tmax) of Emraclidine | Pre-dose and at multiple time points post-dose on Days 1 to 6 in Period 1 and Days 6 to 11 in Period 2
Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-t) of Emraclidine | Pre-dose and at multiple time points post-dose on Days 1 to 6 in Period 1 and Days 6 to 11 in Period 2
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Emraclidine | Pre-dose and at multiple time points post-dose on Days 1 to 6 in Period 1 and Days 6 to 11 in Period 2

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to 29 days
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to 45 days
Number of Participants With Clinically Significant Changes in Vital Sign Parameters | Up to 45 days
Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments | Up to 45 days
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to 45 days
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 45 days
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilworth, Minnesota, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No